CLINICAL TRIAL: NCT04083885
Title: Home-based and Residence-based Virtual Reality Training to Increase Rehabilitative Exercise in Seniors
Brief Title: Virtual Reality Training to Increase Rehabilitative Exercise in Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: York Care Centre (Unknown); Carleton Manor Nursing Home (Unknown); Centre for Innovation and Research in Aging, Canada (Other); Nashwaak Villa (Unknown); Brunswick Hall (Unknown); Loch Lomond Villa (Unknown); Windsor Court Retirement Residence (Unknown); Orchard View Long Term Care Home (Unknown)
Responsible Party: Principal Investigator, Lisa Sheehy, Affiliate Investigator, Bruyère Health Research Institute.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M16-19-026
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Old Age; Debility; Aging
Keywords: rehabilitation; virtual reality; telerehabilitation; technology
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Multi-site Prospective randomized open blinded end-point (PROBE) study
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not know which arm the participants are in. Group allocation will be provided to the research staff member providing the intervention, through use of an online randomization program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants receive 8 weeks of home-based or facility-based virtual reality training, supervised remotely and asynchronously, in addition to their usual activity.
  Interventions: Other: Virtual Reality
- Usual Care (No Intervention): Participants perform their usual activities.

INTERVENTIONS:
Other: Virtual Reality — Participants will be provided with a virtual reality training program, personalized with respect to their abilities, endurance, needs and treatment goals. They will be trained to use the program and it will be installed in their home or provided at their long-term care facility. Participants will be suggested to perform VR 3-5 times a week for 8 weeks. Sessions will be 20-30 minutes long, depending on tolerance.
  Arms: Virtual Reality

SUMMARY:
Seniors are at risk for reduced independence and lowered quality of life after injury or illness. Gains in strength, stamina, balance, cardiovascular fitness and confidence resulting from regular exercise can help seniors to maintain (or improve) their functional ability, independence, and quality of life. However, seniors experience many barriers to exercise. The objective is to assess the use of virtual reality (VR) as a motivating way to encourage seniors to do regular rehabilitative exercise. Seniors who could benefit from rehabilitative exercise and who live in two situations, a) long-term care and b) independently in their homes, will be recruited. Participants will be randomized to usual activity (control) or usual activity plus VR exercise. Long-term care residents will do VR with the assistance of care staff or study partners under the direction of the research team. Independent-living participants will do VR in their homes with the supervision of study partners, under the direction of the research team. All participants will be asked to do VR 3-5 times a week for 8 weeks. Mobility (balance, gait, physical function), and health outcomes (falls, hospital admissions) will be assessed and compared over time.

DETAILED DESCRIPTION:
Background and Justification:

Decreased physical conditioning can occur after injury or illness, particularly in seniors. Frail and physically vulnerable seniors have greater risk for loss of independence and lowered quality of life. They are more likely to need long-term residential care. Seniors also have an increased risk of falls, which are the leading cause of injuries and injury-related hospital admissions among older Canadians, accounting for 85% of seniors' injury-related hospitalizations. Further, falls are associated with over 1/3 of admissions to long-term care facilities after release from the hospital. In 2004, the direct cost of falls to seniors in Canada was estimated to be $2 billion; this number will be much higher today, as health-care costs have increased and the number of seniors has increased as well. Among the many risk factors for falls include physical considerations such as balance and gait deficits, muscle weakness & reduced physical fitness.

Seniors would like to live in their own homes and communities for as long as possible. They also would like to maintain (or improve) their independence, ability to function and quality of life. Gains in strength, stamina, balance, cardiovascular fitness and confidence resulting from regular exercise can help seniors to achieve these goals, reduce the risk of falls and increase social engagement. However, seniors experience many barriers to doing exercise, including a lack of motivation, pain or injury, lack of knowledge, fear of falling, transportation difficulties, no one to exercise with, poor weather and high cost. In fact, only 11% of Canadians between the ages of 60 and 79 meet Canada's physical activity guidelines. For those who live in rural locations, further barriers exist, like isolation, safety (cannot go for a walk on busy highways or dark roads) and lack of access to community-based services.

Virtual reality (VR) is proposed as a motivating and enjoyable way to encourage seniors to do regular rehabilitative exercise, either as part of a home-based rehabilitation plan after injury or illness, or as a part of a plan to enhance mobility and decrease falls in a residential long-term care home.

Goals:

1. To assess the impact of adding home-based VR exercise to usual activity of community-based residents.
2. To assess the impact of adding facility-based VR exercise to usual activity of residents living in long-term care.

Objectives:

1. To assess the impact of 8 weeks of home-based VR as an addition to usual activity on:

   1. balance, physical function, community integration and quality of life;
   2. number of falls, number of emergency room visits, hospital admissions and long-term care admissions;
   3. acceptance of VR for exercise.
2. To assess the impact of 8 weeks of facility-based VR as an addition to usual activity of residents in long-term care on:

   1. balance, physical function and quality of life;
   2. number of falls, number of emergency room visits, hospital admissions;
   3. acceptance of VR for exercise.

Two separate, but related studies are included; A) Randomized controlled trial studying the addition of home-based VR to usual activity, compared to usual activity only, for participants living independently in their homes.

B) Multi-site randomized controlled trial studying the addition of facility-based VR to usual activity, compared to usual activity only for participants living in long-term care facilities.

A) Home-based study participants will undergo a 1-1 1/2 hour physical assessment of balance, gait, physical function, activities of daily living and quality of life, given by the Research Assistant (RA), either in their homes or at the Centre for Innovation and Research on Aging (CIRA). The Research Therapist (RT) will assess the participant's 5 m walk test (used to assess gait speed; Appendix U), then randomize the participant into either the control or experimental groups using an online randomization tool, stratified according to gait speed.

Participants in the control group will be told to continue on as normal with their usual activities.

Participants and study partners in the experimental group will be introduced to the Jintronix VR platform and will discuss with the RT their abilities and therapy goals. The RT will consult with the participant's health care professionals (if appropriate) and create a customized VR program of approximately 20-30 minutes. The RT will then install the VR system in the participant's home and train the participant and study partner on the use of VR. Safety considerations will be reviewed (the study partner is not to assist or guard the participant, just be in the home during VR). A photograph is taken of the set-up, to document that the location is safe, in case the participant re-arranges furniture etc. into an unsafe position.

Participants will be instructed to perform the VR session 3-5 times a week for 8 weeks. The RT will contact the participant (preferably by phone) twice in the first week and at least once a week thereafter, and participants will be invited to contact the RT as needed. The RT will also monitor VR usage remotely. The RT can modify the games remotely as required. Further home visits can be made as required, preferably once during week 2, to assess exercise technique and answer questions.

After 8 weeks, the participant will return to CIRA to be reassessed by the RA and then the VR system will be removed from the home. The first 10 participants in the experimental group (and their study partners) will also provide a 10-minute interview on their experience with VR.

One month later, the participant will return to CIRA for a final reassessment with the RA.

All assessments can be performed in the participant's home rather than having them come to CIRA.

B) Facility-based study participants will undergo a 1 - 1 ½ hour physical assessment of balance, gait, physical function, activities of daily living and quality of life, given by the Research Assistant (RA). This assessment will be done at the participant's long-term care facility. The Research Therapist (RT) will assess the participant's 5 m walk test (used to assess gait speed; Appendix U), then randomize the participant into either the control or experimental groups using an online randomization tool, stratified according to gait speed.

Participants in the control group will be told to continue on as normal with their Extra-Mural homecare rehabilitation program and/or any other activities that they normally do.

Participants in the experimental group will be introduced to the Jintronix VR platform and will discuss with the RT their abilities and therapy goals. The RT will consult with the participant's health care professionals (if appropriate) and with the facility staff (particularly recreation therapists and rehabilitation assistants), and create a customized VR program of approximately 20-30 minutes.

Rehabilitation assistants and recreation therapists/coordinators working at the long-term care sites will be trained on the use of Jintronix VR during a 2-hour workshop. The rehabilitation assistants or recreation therapists/coordinators will be instructed on each participant's individual program and any safety or technique requirements and will assist and supervise long-term care participants to perform their VR programs. Other study partners (for example, family members or volunteers) may be used as well. Participants will be instructed to perform the VR session 3-5 times a week for 8 weeks. The RT will contact the participant and the rehabilitation assistant or recreation therapist or study partner (preferably in person) twice in the first week and at least once a week thereafter, and participants and rehabilitation assistant/recreation therapist/study partner will be invited to contact the RT as needed. The RT will also monitor VR usage remotely. The RT can modify the games remotely as required.

After 8 weeks, all participants will be reassessed at their long-term care facilities by the RA. The first 10 residents in the experimental group will also provide a 10-minute interview on their experience with VR. One month later, the participant will have a final reassessment with the RA.

ELIGIBILITY:
Inclusion Criteria:

Home-based VR - Eligible are seniors (=> 65 years old) with reduced mobility or functional decline, or who could benefit from increased rehabilitative exercise. Clients must 1) be able to sit or stand without assist (gait aid is fine) for 20 minutes (rest breaks are fine), 2) have sufficient cognitive ability to perform VR, 3) have a study partner, 4) speak and understand French or English, 5) attend 3 sessions at the assessment site or their own home, 6) have enough space in their home, 7) have no health conditions that preclude mild to moderate exercise, 8) live within 50km of the assessment site.

Facility-based VR - Eligible are seniors living in long-term care and receiving rehabilitation or maintenance programs for mobility issues or functional decline, or who could benefit from rehabilitative exercise. Residents must 1) be able to sit or stand without assist (gait aid is fine) for at least 20 minutes (rest breaks are fine), 2) have sufficient cognitive ability to perform VR, 3) speak and understand French or English, 4) have no health conditions that preclude mild exercise, 5) have a study partner (can be a staff member, family member, friend, volunteer etc.).

Exclusion Criteria:

Patients will be excluded if they have an unstable medical condition, seizures or vertigo.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Functional Reach Test | Change from baseline to immediately after 8-week intervention
  Measures stability by measuring the maximum distance one can reach forward. Longer distance is better.

SECONDARY OUTCOMES:
Functional Reach Test | Change from immediately after 8-week intervention to 1 month later
  Measures stability by measuring the maximum distance one can reach forward. Longer distance is better.
Berg Balance Scale | Change from baseline to immediately after 8-week intervention
  Measures standing balance and physical function;14 items scored from 0-4 summed for a total out of 56 (higher is better)
Berg Balance Scale | Change from immediately after 8-week intervention to 1 month later
  Measures standing balance and physical function;14 items scored from 0-4 summed for a total out of 56 (higher is better)
Timed Up and Go | Change from baseline to immediately after 8-week intervention
  Measures the time required to rise from a chair, walk 3 m, return and sit down (3 versions, original, manual (carrying a cup of water) and cognitive (count backward in 3's from 99)) Lower time is better.
Timed Up and Go | Change from immediately after 8-week intervention to 1 month later
  Measures the time required to rise from a chair, walk 3 m, return and sit down (3 versions, original, manual (carrying a cup of water) and cognitive (count backward in 3's from 99)) Lower time is better.
Five Times Sit to Stand | Change from baseline to immediately after 8-week intervention
  Measures lower extremity strength by timing how long it takes to stand then sit 5 times. Lower time better.
Five Times Sit to Stand | Change from immediately after 8-week intervention to 1 month later
  Measures lower extremity strength by timing how long it takes to stand then sit 5 times. Lower time better.
Frenchay Activities Index | Change from baseline to immediately after 8-week intervention
  Measures the frequency of domestic chores, leisure/work and outdoor activities. Scores 15 items from 0-3, summed for a total score out of 45. Higher is better.
Frenchay Activities Index | Change from immediately after 8-week intervention to 1 month later
  Measures the frequency of domestic chores, leisure/work and outdoor activities. Scores 15 items from 0-3, summed for a total score out of 45. Higher is better.
Medical Outcomes Study Short Form 36 (SF-36) | Change from baseline to immediately after 8-week intervention
  Patient report of health status and health-related quality of life. Rates 36 items from 1-3, 1-2, 1-5 or 1-6 and uses "rules" to score each out of 100 and averages them in groups to create scores in 8 different categories (ex. energy/fatigue, emotional well-being). Higher is better.
Medical Outcomes Study Short Form 36 (SF-36) | Change from immediately after 8-week intervention to 1 month later
  Patient report of health status and health-related quality of life. Rates 36 items from 1-3, 1-2, 1-5 or 1-6 and uses "rules" to score each out of 100 and averages them in groups to create scores in 8 different categories (ex. energy/fatigue, emotional well-being). Higher is better.
Feasibility of Virtual Reality | Immediately after 8-week intervention
  Semi-structured Participant and Study Partner Questionnaire interview on enjoyment, perceived usefulness and acceptance of virtual reality, and interest to continue using VR.
Falls | Measured during 8-week intervention
  Number of falls
Falls | Measured during 1-month post-intervention phase
  Number of falls
Emergency Room Visits | Measured during 8-week intervention
  Number of emergency room visits
Emergency Room Visits | Measured during 1-month post-intervention phase
  Number of emergency room visits
Hospital Admissions | Measured during 8-week intervention
  Number of admissions to hospital
Hospital Admissions | Measured during 1-month post-intervention phase
  Number of admissions to hospital
Long-term Care Admissions | Measured during 8-week intervention
  Number of admissions to long-term care
Long-term Care Admissions | Measured during 1-month post-intervention phase
  Number of admissions to long-term care
Utilization of Virtual Reality - Days | Measured during 8-week intervention
  Number of days VR was used
Utilization of Virtual Reality - Minutes | Measured during 8-week intervention
  Average number of minutes VR was used during each session

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Sheehy, PhD, Principal Investigator — Bruyère Health Research Institute.; Justine Henry, MSc, Principal Investigator — Centre for Innovation and Research in Aging, Canada
Locations (7):
- Canada (7):
  - York Care Centre, Fredericton, New Brunswick
  - Windsor Court, Fredericton, New Brunswick
  - Brunswick Hall Special Care Home, Fredericton, New Brunswick
  - Orchard View Long Term Care Home, Gagetown, New Brunswick
  - Loch Lomond Villa, Saint John, New Brunswick
  - Nashwaak Villa, Stanley, New Brunswick
  - Carleton Manor Nursing Home, Woodstock, New Brunswick

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheehy L, Taillon-Hobson A, Sveistrup H, Bilodeau M, Yang C, Welch V, Hossain A, Finestone H. Home-based virtual reality training after discharge from hospital-based stroke rehabilitation: a parallel randomized feasibility trial. Trials. 2019 Jun 7;20(1):333. doi: 10.1186/s13063-019-3438-9. PMID 31174579
- [Result] Sheehy L, Chapman I, Sveistrup H, Yang C, Bilodeau M, Finestone H. Home-based virtual reality training after stroke: preliminary data of a telerehabilitation feasibility randomized controlled trial. International Journal of Stroke 13(2S):207, 2018.
- [Derived] Sheehy L, Bharadwaj L, Nissen KA, Estey JL. Non-Immersive Virtual Reality Exercise Can Increase Exercise in Older Adults Living in the Community and in Long-Term Care: A Randomized Controlled Trial. Clin Interv Aging. 2025 Feb 5;20:109-124. doi: 10.2147/CIA.S498272. eCollection 2025. PMID 39931102
- See also: Bruyere Research Institute — https://www.bruyere.org/en/about-bri
- See also: Centre for Innovation and Research in Aging — https://agingresearch.ca/